CLINICAL TRIAL: NCT00046020
Title: An Acute and Continuation Phase Study of the Comparative Efficacy Study of Venlafaxine ER (Effexor® XR) and Fluoxetine (Prozac®) in Achieving and Sustaining Remission (Wellness) in Patients With Recurrent Unipolar Major Depression; Followed by a Long Term Randomized, Placebo-Controlled Maintenance Treatment Study in Patients Treated Initially With Venlafaxine ER
Brief Title: Study Evaluating Venlafaxine ER in Recurrent Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Purpose: Treatment
Other Study IDs: 0600B-100469
Record Dates: First submitted 2002-09-18; First posted 2002-09-19 (Estimated); Last update posted 2009-08-14 (Estimated); Status verified 2009-08

CONDITIONS: Depressive Disorder, Major; Recurrence
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence; Depression

INTERVENTIONS:
Drug: Venlafaxine ER

SUMMARY:
The purpose of this study is to review the long-term comparative efficacy of venlafaxine ER in achieving and sustaining remission (wellness) in patients with recurrent major depression

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis for recurrent major depression

Exclusion Criteria

* The patient has failed on an adequate trial of fluoxetine, venlafaxine or venlafaxine ER during the current episode of major depression or the patient is treatment-resistant
* Known hypersensitivity to venlafaxine or fluoxetine
* History or presence of clinically significant hepatic, cardiovascular or renal disease, or other serious medical disease, including history of seizure disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1096 (Actual)
Dates: Start 2000-08; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Kornstein SG, Pedersen RD, Holland PJ, Nemeroff CB, Rothschild AJ, Thase ME, Trivedi MH, Ninan PT, Keller MB. Influence of sex and menopausal status on response, remission, and recurrence in patients with recurrent major depressive disorder treated with venlafaxine extended release or fluoxetine: analysis of data from the PREVENT study. J Clin Psychiatry. 2014 Jan;75(1):62-8. doi: 10.4088/JCP.12m07841. PMID 24345717
- [Derived] Keller MB, Trivedi MH, Thase ME, Shelton RC, Kornstein SG, Nemeroff CB, Friedman ES, Gelenberg AJ, Kocsis JH, Dunner DL, Hirschfeld RM, Rothschild AJ, Ferguson JM, Schatzberg AF, Zajecka JM, Pedersen RD, Yan B, Ahmed S, Musgnung J, Ninan PT. The Prevention of Recurrent Episodes of Depression with Venlafaxine for Two Years (PREVENT) Study: Outcomes from the 2-year and combined maintenance phases. J Clin Psychiatry. 2007 Aug;68(8):1246-56. doi: 10.4088/jcp.v68n0812. PMID 17854250
- [Derived] Kocsis JH, Thase ME, Trivedi MH, Shelton RC, Kornstein SG, Nemeroff CB, Friedman ES, Gelenberg AJ, Dunner DL, Hirschfeld RM, Rothschild AJ, Ferguson JM, Schatzberg AF, Zajecka JM, Pedersen RD, Yan B, Ahmed S, Musgnung J, Ninan PT, Keller MB. Prevention of recurrent episodes of depression with venlafaxine ER in a 1-year maintenance phase from the PREVENT Study. J Clin Psychiatry. 2007 Jul;68(7):1014-23. doi: 10.4088/jcp.v68n0706. PMID 17685736